CLINICAL TRIAL: NCT05472558
Title: Clinical Study of Cord Blood-derived CAR-NK Cells Targeting CD19 in the Treatment of Refractory/Relapsed B-cell NHL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0496
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB CAR-NK019 (Experimental): All subjects were intravenously administrated with CAR-NK019
  Interventions: Biological: anti-CD19 CAR-NK

INTERVENTIONS:
Biological: anti-CD19 CAR-NK — lentiviral vector-transducted cord blood-derived NK cells to express anti-CD19 CAR
  Other Names: CB CAR-NK019

SUMMARY:
To study the safety and effectiveness of cord blood-derived CAR-NK cells targeting CD19 in patients with B-cell non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
This is an open, single-arm, single-dose, dose-escalation clinical trial designed to evaluate the safety and the preliminary efficacy of CB CAR-NK019 cells. 9-18 patients are planned to be enrolled in the dose-escalation trial (2×10^6 cells/kg ,3×10^6 cells/kg, 4×10^6 cells/kg) . The primary endpoints are DLT, MTD, and the second endpionts are the overall response rates (CR and PR), overall survival, and progression-free survival. Based on the results in the dose-escalation trial, the recommended dose will be determined. Another 30 patients will be enrolled to estimate the safety and efficacy of CB CAR-NK019 under the best dose.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Volunteer to participate in this study and sign an informed consent form; Age 18-75 years old, no gender limit;

Histologically diagnosed as diffuse large B-cell lymphoma (DLBCL), transforming follicular lymphoma (TFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL) and other inert B-cells NHL conversion type:

Refractory or relapsed DLBCL refers to the failure to achieve complete remission after 2-line treatment; disease progression during any treatment, or disease stable time equal to or less than 6 months; or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation ； Refractory or relapsed MCL must be resistant to or intolerable to BTK inhibitors; Refractory or relapsed indolent B-cell NHL is the failure or recurrence of third-line treatment; Previous treatment must include CD20 monoclonal antibody treatment (unless the subject is CD20 negative) and anthracyclines; At least one measurable lesion with the longest diameter ≥ 1.5 cm exists; The expected survival period is ≥12 weeks; The puncture section of the tumor tissue was positive for CD19 expression; ECOG score 0-2 points;

Sufficient organ function reserve:

Alanine aminotransferase, aspartate aminotransferase ≤ 2.5× UNL (upper limit of normal value); Creatinine clearance rate (Cockcroft-Gault method) ≥60 mL/min; Serum total bilirubin and alkaline phosphatase ≤1.5× UNL; Glomerular filtration rate>50Ml/min Cardiac ejection fraction (EF) ≥50%; Under natural indoor air environment, basic oxygen saturation>92% Allow a previous stem cell transplantation The approved anti-B-cell lymphoma treatments, such as systemic chemotherapy, systemic radiotherapy, and immunotherapy, have been completed for at least 3 weeks before the study medication; Allow patients who have previously received CAR-T cell therapy and have failed or relapsed after 3 months of evaluation; Female subjects of childbearing age must have a negative pregnancy test and agree to take effective contraceptive measures during the trial Two tests for the new coronavirus were negative.

Exclusion Criteria:

* Those who have a history of allergies to any of the ingredients in cell products; History of other tumors Previously presented with II-IV degree (Glucksberg criteria) acute GvHD or extensive chronic GvHD; or are receiving anti-GvHD treatment; Have received gene therapy in the past 3 months; Active infections that require treatment (except for simple urinary tract infections and bacterial pharyngitis), but preventive antibiotics, antiviral and antifungal infection treatments are allowed; Hepatitis B (HBsAg positive, but HBV-DNA <103 is not an exclusion criterion) or hepatitis C virus infection (including virus carriers), syphilis and other subjects with acquired and congenital immunodeficiency diseases, including But not limited to people living with HIV; According to the New York Heart Association's Heart Function Classification Standard, it is classified as Grade III or Grade IV.

Impaired subjects;

Those who have received anti-tumor therapy in the early stage but the toxic reaction has not recovered (the CTCAE 5.0 toxic reaction has not recovered to ≤1, except for fatigue, anorexia, and hair loss); Subjects with a history of epilepsy or other central nervous system diseases; Enhanced CT or MRI of the head showed evidence of central nervous system lymphoma; Have received any other drugs that target CD19; Women who are breastfeeding and unwilling to stop breastfeeding; Any other situation that the investigator believes may increase the risk of the subject or interfere with the results of the test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of cord blood-derived Anti-CD19 CAR-NK Cell Therapy for B-cell Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
Complete response rate (CR) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Duration of response (DOR) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Partial response rate (PR) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Overall response rate (ORR) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Immunogenicity after the infusion of CB CAR-NK019 | Up to 2 years
  To evaluate the immunogenicity of CB CAR-NK019

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No